CLINICAL TRIAL: NCT04280302
Title: Realitat Virtual Com a Tractament Coadjuvant en rehabilitació Vestibular
Brief Title: Virtual Reality-based Rehabilitation
Acronym: VRVEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Pompeu Fabra (Other)
Responsible Party: Principal Investigator, Paul Verschure, PhD, Universitat Pompeu Fabra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VESTHJXXIII
Record Dates: First submitted 2020-02-14; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Patients With Unilateral Peripheral Vestibular Deficits
Keywords: vestibular; unilateral vestibular; virtual reality; rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality based therapy (Experimental)
  Interventions: Behavioral: Virtual Reality-based Rehabilitation
- Conventional Therapy (Active Comparator)
  Interventions: Behavioral: Conventional Therapy

INTERVENTIONS:
Behavioral: Virtual Reality-based Rehabilitation — VR-based eye stabilization exercises and balance exercises
  Arms: Virtual reality based therapy
Behavioral: Conventional Therapy — Conventional rehabilitation therapy based on eye stabilization exercises and balance exercises
  Arms: Conventional Therapy

SUMMARY:
Vertigo / dizziness, imbalance and other symptoms related to vestibular pathology have a life prevalence of 7.4%. Peripheral and unilateral vestibulopathy are among the most common types, and in some patients the symptoms become chronic and disabling, which makes it difficult for them to lead a normal life and has a significant socio-economic impact. In recent years, the effect of vestibular rehabilitation with virtual reality has been studied and positive results have been obtained when compared with traditional rehabilitation, but despite rehabilitation there is patients who are still chronic, and the reasons for this prognostic variability are still unknown and require further treatment. Virtual reality-based stimulation can play a significant role as an adjunct to conventional vestibular rehabilitation, improving its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral vestibular deficit
* Vestibular neuritis
* Sudden hearing loss with vestibular involvement
* Labyrinthitis
* Ménière's disease
* Vestibular Shwannoma
* Benign paroxysmal positional vertigo
* Vestibular symptoms (vertigo, dizziness, imbalance, gait instability, kinosis and / or oscillopsy) chronic (more than 6 weeks of evolution)
* Over 18 years old

Exclusion Criteria:

* Failure to meet some of the inclusion criteria
* Neurological, traumatological, rheumatological, ophthalmological or systemic pathology that may interfere with the balance
* Inability to understand participation in the study
* Non-acceptance to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Change pre-post treatment in the Dizziness handicap inventory (DHI) (0-100) | 4 weeks
  Change within subjects from baseline to the end of week 4

SECONDARY OUTCOMES:
Change pre-post treatment in Posturography (Wii+software RombergLab) | 4 weeks
  Change within subjects from baseline to the end of week 4
Change pre-post treatment in Test up and go (TUG) | 4 weeks
  Change within subjects from baseline to the end of week 4
Change pre-post treatment in Berg Scale (0-56) | 4 weeks
  Change within subjects from baseline to the end of week 4
Change pre-post treatment in Tinneti Test (1-28) | 4 weeks
  Change within subjects from baseline to the end of week 4
Change pre-post treatment in Simulator Sickness Questionnaire (SSQ) (0-14) | 4 weeks
  Change within subjects from baseline to the end of week 4
Change pre-post treatment in the Video-head impulse test (vHIT) | 4 weeks
  Change within subjects from baseline to the end of week 4
Change pre-post treatment in the Barthel Index (0-100) | 4 weeks
  Change within subjects from baseline to the end of week 4
Change pre-post treatment in the SF 12 Test (0-100) | 4 weeks
  Change within subjects from baseline to the end of week 4

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Sáez Felipe, Principal Investigator — ssaezfelipe@gmail.com
Locations (1):
- Hospital Universitari de Tarragona Joan XXIII, Tarragona, Spain